CLINICAL TRIAL: NCT03201315
Title: The Incremental Risk of Intraoperative Fentanyl on PONV: A Modifiable Risk Without Drawbacks?
Brief Title: The Incremental Risk of Intraoperative Fentanyl on PONV
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2016-01605
Record Dates: First submitted 2017-05-17; First posted 2017-06-28 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: PONV
Keywords: Fentanyl, opioids
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this quality control study is to describe the presence and intensity of postoperative nausea and vomiting (PONV) and its correlation with intraoperative fentanyl dosing. Additionally, the investigators will examine pain scores.

DETAILED DESCRIPTION:
The primary aims of this quality control study are:

1. to determine whether there is an independent association between the intraoperative administration of fentanyl (both as a continuous and categorical variable) and PONV within 24 postoperative hours
2. determine whether or not the intraoperative fentanyl amount can be used to successfully restratify patients for PONV beyond the simplified Apfel score for PONV

All required data is collected in regular daily practice. The following variables will be assessed by univariable models:

Preoperative variables (e.g. patient characteristics) Surgical/Anesthesia variables (e.g. type/length of surgery, antiemetics) Outcome variables (PONV, worst pain as delineated in the outcomes section), Intraoperative fentanyl measured 1) as a continuous variable and 2) by predefined limits of 0 to 0.2mg, >0.2-0.5mg, >0.5 to 0.8mg, and >8mg.

Finally for the multivariable model, the investigators will adjust for confounders, specifically for sex (m/f), history (Hx) of PONV (y/n), Hx of motion sickness (y/n), current smoker (y/n), age (years), expected duration of surgery (min; >60 min), postoperative opioids (y/n), the use of preemptive PONV Therapy (0,1,2 medications), propofol vs. inhalative agents (y/n), and surgery type (3 kinds) from the patient's electronic record. In the event that insufficient event rates are observed, we will collapse the variables into the simplified Apfel score to assess the independent value of fentanyl in predicting PONV.

In addition to a logistic model as delineated above, we will conduct the following:

1. receiver operating characteristic (ROC) curves of the logistic model without fentanyl, with fentanyl (continuous), and with fentanyl (categorical).
2. additionally, ROCs of a simplified model using the Apfel score, the Apfel score with fentanyl (continous), and the Apfel score with fentanyl (categorical) will be made. Comparison of area under the receiver operating characteristics(AUROCs) by DeLong
3. net reclassification improvement (NRI) of both the logistic model with and without fentanyl as well as the Apfel score with and without fentanyl

To assess pain and administered fentanyl, we will examine pain scores by the numeric rating scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* In-patients with an expected simplified Apfel score of 2 or higher,
* Aged >= 18 years, and
* Undergoing general anesthesia (with or without neuraxial or regional anesthesia.)
* in abdominal, gynecological or otorhinolaryngological surgery

Exclusion Criteria:

* Outpatients
* Patients with chronic pain, defined as recurring pain requiring intermittent hospitalization or regular intake of pain medication.
* Non-opioid naïve patients, defined as a history of abuse or having taken opioids within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an elevated PONV risk undergoing abdominal, gynecological, or otorhinolaryngological in-patient surgery
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Any postoperative nausea and/or vomiting (PONV) within 24 hours after surgery | within 24 hours (or next morning discharge)
  postoperative nausea and/or vomiting (PONV) yes/no (either by chart or by patient confirmation) within 24 hours (or next morning discharge)

SECONDARY OUTCOMES:
number of postoperative vomiting events within 24 hours | within 24 hours (or next morning discharge)
  Number of times vomiting (0, 1-2, >3 times; either by chart or by patient confirmation) within 24 hours (or next morning discharge)
Any postoperative nausea and/or vomiting (PONV) while in the recovery room | first two postoperative hours
  Postoperative nausea and/or vomiting (PONV) yes/no (either by chart or by patient confirmation) while in recovery room
Worst pain, i.e. highest Numeric Rating Score (NRS) | within 24 hours / in recovery room (first two postoperative hours)
  highest / worst pain score within 24 hours / in recovery room (defined as above)

OTHER OUTCOMES:
Dose of postoperative administration of opioids | within 24 hours / in recovery room (first two postoperative hours)
  quantification of postoperative administration of opioids 24 hours/recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Bandschapp, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland; Wilhelm Ruppen, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland; Eckhard Mauermann, MD, MSc, Principal Investigator — University Hospital Basel; University Hospital Ghent
Locations (1):
- Universitiy Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mauermann E, Clamer D, Ruppen W, Bandschapp O. Association between intra-operative fentanyl dosing and postoperative nausea/vomiting and pain: A prospective cohort study. Eur J Anaesthesiol. 2019 Nov;36(11):871-880. doi: 10.1097/EJA.0000000000001081. PMID 31567573